CLINICAL TRIAL: NCT06321497
Title: Measuring the Impact of Extracorporeal Carbon Dioxide Removal Using PrismaLung in Reducing Ventilator Induced Lung Injury in Mechanically Ventilated Patients
Brief Title: Extracorporeal Carbon Dioxide Removal Using PrismaLung in Reducing Ventilator Induced Lung Injury
Status: Recruiting | Type: Observational
Sponsor: Peninsula Health (Other Government)
Collaborators: Monash University (Other); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 85711
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2023-12

CONDITIONS: ARDS, Human
Keywords: ECC2R, Carbon dioxide, ventilator induced lung injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients (18 years or older) with diagnosis of ARDS as per Berlin Definition
  Interventions: Device: Extracorporeal carbon dioxide removal

INTERVENTIONS:
Device: Extracorporeal carbon dioxide removal — Low flow extracorporeal carbon dioxide removal with PrismaLung+

SUMMARY:
Lung protective ventilation with low tidal volumes and low driving pressure are known to reduce mortality in mechanically ventilated patients with acute respiratory failure. This reduction in mortality is known be due to reduction of ventilator induced lung injury that occurs due to high tidal volumes and high driving pressure. When receiving such mechanical ventilation, some patients develop hypercapnia and associated hypercapnic acidosis. Such patients have an increased risk of mortality. While the exact reasons for such increase in mortality is not known, it is recommended to minimise hypercapnia and hypercapnic acidosis during lung protective ventilation. Minimally invasive extracorporeal carbon dioxide removal (ECCO2R) devices are shown to reduce hypercapnia and hypercapnic acidosis. There are several devices that are currently available in the current clinical practice. However, the effect of these devices on reduction in ventilator induced lung injury is not clearly demonstrated. This study aims to assess the use of an ECCO2R device called Prismalung in reducing ventilator induced lung injury. PrismaLung is currently used in our intensive care unit. This assessment is done by measuring interleukins in bronchoalveolar lavage fluid and blood interleukin levels as well as clinical assessment including the reduction of driving pressure.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (18 years or older) with diagnosis of ARDS as per Berlin Definition21.

Driving pressure (ΔP) > 14 and/or Plateau >/= 25 (ΔP is calculated using as plateau pressure minus positive end-expiratory pressure)20 Respiratory rate > 20 breaths per minute pH < 7.25 and PaCO2 >45

Exclusion Criteria:

ARDS lasting more than 72 hours at the time of inclusion High pressure (Plateau pressure >30 cm H2O) or high FiO2 (>0·8) ventilation for more than 168 h (7 days); Life threatening hemodynamic instability as defined by ongoing arrhythmias that is not responsive to treatment Contraindication to limited anticoagulation Treatment limitation including not for resuscitation and not for reintubation Patients with potentially irreversible respiratory failure caused by conditions such as pulmonary fibrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18 years or older) with diagnosis of ARDS
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Reduction in driving airway pressures | 72 and 144 hours post initiation of ECCO2R

SECONDARY OUTCOMES:
Reduction in pulmonary inflammation assessed by interleukins in lung | 72 and 144 hours post initiation of ECCO2R

CONTACTS AND LOCATIONS:
Overall Officials: RAVINDRANATH TIRUVOIPATI, PhD, Principal Investigator — Peninsula Heatlh
Locations (1):
- Frankston Hospital, Frankston, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No